CLINICAL TRIAL: NCT05191394
Title: IMPACT OF THERAPEUTIC PLASMA EXCHANGE ON ACQUIRED VACCINAL ANTI-SARS-CoV-2 ANTIBODIES.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/08SEP/367
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Therapeutic Plasma Exchange
Keywords: Therapeutic plasma exchange; anti-SARS-CoV-2 antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evolution of anti-SARS-CoV-2 titer over time in vaccinated adult patients treated with TPE. (Other): Assessment of the possible variation of anti-SARS-CoV-2 antibody titer in adult patients regularly treated with therapeutic plasma exchange.
  For each patient included in this study, 3 blood samples of 5 ml(serum) will be collected at well-defined time points: at the beginning of an TPE session, at the end of the same session, and at the beginning of the consecutive TPE session.
  Interventions: Diagnostic Test: Evolution of antibodies titre

INTERVENTIONS:
Diagnostic Test: Evolution of antibodies titre — For each patient included in this study, 3 blood samples of 5 ml(serum) will be collected at well-defined time points: at the beginning of an TPE session, at the end of the same session, and at the beginning of the consecutive TPE session.

SUMMARY:
Context:

Therapeutic plasma exchange is an extracorporeal blood purification technique that removes pathogenic substances (including antibodies) from plasma. This technique also combines an immunomodulatory effect. The impact on the anti-SARS-CoV-2 titre and the humoral and cellular responses in the general population benefiting from therapeutic plasma exchanges is not known at this time.

The purpose of this study is to evaluate the evolution of anti-SARS-CoV-2 antibodies' titre over time in vaccinated adult patients treated with therapeutic plasma exchange.

Research question and associated variables:

Prospective non-drug interventional study on the possible variation of anti-SARS-CoV-2 antibody titre in adult patients regularly treated with therapeutic plasma exchange.

Study population: any adult patient vaccinated against SARS-CoV-2 (any type of vaccine) and regularly receiving therapeutic plasma exchange in the adult hematology department of the Cliniques universitaires Saint Luc in Brussels, Belgium.

Number of subjects expected to be enrolled: 10-15

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Adult patients vaccinated against SARS-CoV-2 (any type of vaccine) and regularly receiving therapeutic plasma exchange in the adult hematology department of the Cliniques universitaires Saint Luc.

Exclusion Criteria:

* Patients treated with therapeutic plasma exchange for an acute condition at the intensive care unit
* Patients unable to sign the ICF or unwilling to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the variation of the anti-SARS-CoV-2 antibodies with plasma exchange procedures | 3 months
  Evolution of anti-SARS-CoV-2 antibodies titre over time in vaccinated adult patients treated with TPE.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lambert, Pr, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, International, Belgium